CLINICAL TRIAL: NCT01180036
Title: "A Randomized Controlled Trial of Rituximab Versus Cyclosporine in the Treatment of Idiopathic Membranous Nephropathy (IMN)"
Brief Title: MEmbranous Nephropathy Trial Of Rituximab
Acronym: MENTOR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Columbia University (Other); University of British Columbia (Other); Ohio State University (Other); Stanford University (Other); University of Washington (Other); University of Michigan (Other); University of Alabama at Birmingham (Other); Case Western Reserve University (Other); The Cleveland Clinic (Other); University of Kansas Medical Center (Other); University of Manchester (Other); University Health Network, Toronto (Other); University of Toronto (Other); CHU de Quebec-Universite Laval (Other); Washington University School of Medicine (Other); Florida International University (Other); University of Mississippi Medical Center (Other); NYU Langone Health (Other); Medical College of Wisconsin (Other); University of Arizona (Other); Sunnybrook Health Sciences Centre (Other); Applied Health Research Centre (Other); Fulk Family Foundation (Unknown)
Responsible Party: Principal Investigator, Fernando Fervenza, M.D., Ph.D, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-003372
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Rituximab; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab Treatment Arm (Active Comparator): Patients randomized to the RTX arm will receive 1000 mg IV on Days 1 and 15. Patients who achieve complete remission at 6 months will not be retreated. A second course of RTX 1000 mg IV will be administered at study month 6 for individuals who have not achieved a complete remission, but have achieved a minimum of >25% reduction in Time 0 proteinuria. Dosing at study month 6 will be independent of cluster of differentiation (CD) 19+ B cell count.
  Interventions: Drug: Rituximab
- Cyclosporine Treatment Arm (Active Comparator): Patients randomized to the Cyclosporine arm will be started at a dose of CsA = 3.5 mg/kg/day p.o. divided into 2 equal doses given at 12 hour intervals. Target trough CsA blood levels are 125 to 175 ng/ml. Patients will have their doses adjusted according to their blood levels of CSA as monitored every 2 weeks until the target trough level is reached. If a complete remission is achieved by 6 months, CSA will be tapered and discontinued over a three-month period. If after 6 months there has not been a reduction in proteinuria of at least 25% of baseline values, the drug will also be discontinued. If there has been a >25% reduction in baseline proteinuria (but not complete remission) the CSA will be continued for an additional 6 months.
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Rituximab — 1000 mg, I.V. on Days 1 and 15 and will be retreated at month 6 independent of cluster of differentiation (CD) 19+ B cell count
  Other Names: Rituxan, MabThera
  Arms: Rituximab Treatment Arm
Drug: Cyclosporine — Patients randomized to the Cyclosporine arm will be started at a dose of (CsA = 3.5 mg/kg/day p.o. divided into 2 doses for 12 months). Target trough CsA blood levels, as determined in whole blood by High Performance Liquid Chromatography (HPLC), are 125 to 175 ng/ml. A persistent and otherwise unexplained increase in serum creatinine >30% would prompt an approximate 25% dose reduction of CSA, aiming for a corresponding 25% reduction in CSA trough level. If with this dose reduction the creatinine does not return to within 30% of baseline levels within 3 weeks, then a second dose reduction of approximately 25% with similar reduction in CSA trough level will be used. If the creatinine does not fall to baseline values with this second dose reduction, the drug will be discontinued. At the end of 12 months, Cyclosporine will be tapered by 1/3 of the maintenance dose monthly and hence discontinued after 3 months.
  Other Names: Sandimmune
  Arms: Cyclosporine Treatment Arm

SUMMARY:
The primary outcome of this study is to determine whether or not the B cell targeting with Rituximab is non-inferior or more effective than Cyclosporine in inducing long term remission of proteinuria.

DETAILED DESCRIPTION:
In IMN, experimental data suggests that B cells are involved in the pathogenesis of the disease. To date, the best proven therapy for patients with MN consists of the combined use of corticosteroids and cyclophosphamide (CYC). Since the mechanism of action of CYC includes suppression of various stages of the B cell cycle including B cell activation, proliferation, and differentiation and inhibition of immunoglobulin (IgG) secretion, it lends credence to the hypothesis that B cells abnormalities are involved in the pathogenesis of MN. Given the key role of IgG antibodies in MN, it is reasonable to postulate that suppression of antibody production by depleting B cells may improve or even resolve the glomerular pathology and be reflected by a reduction in proteinuria. Thus, a case could be made for using an agent capable of selectively depleting B cells, and therefore halting the production of immunoglobulins against antigens potentially present in the glomeruli. This approach could stop the initiating sequence of pathogenic events and result in resolution of the. The P.I. believes that the application of selective B cell targeting with Rituximab (RTX) will prove at least equal, or even superior, both in the production of short term and long term control of the nephrotic syndrome (NS) and be safer than any current therapeutic regimen used to treat MN.

Based on this rationale, the investigators conducted a pilot trial in 15 newly-biopsied patients (<3 years) with IMN and proteinuria >5g/24h despite ACEi/ARB use for >3months and systolic BP <130 millimeter of mercury (mmHg). Mean baseline creatinine was 1.4 mg/dl. Thirteen males and 2 females, median age 47 (range 33-63), were treated with RTX (1g) on days 1 and 15. At six months, patients who remained with proteinuria >3g/24 received a second identical course of RTX. Baseline proteinuria of 13.0±5.7g/24h (range 8.4-23.5) decreased to 6.0±7.0 g/24h (range 0.2-20) at 12 months (mean ± SD). In the fourteen patients who completed a 12 months follow-up complete remission (proteinuria <0.3g/24h) was achieved in 2 patients and partial remission (<3g/24h) in 7 patients. In 5 of these 7 patients, proteinuria was <1.5g/24h and follow up at 18 months showed that 3 of these 7 patients on PR achieved CR of proteinuria. Five patients did not respond. The mean drop in proteinuria from baseline to 12 months was 6.2± 5.1g (p=.002, paired t-test). There were a limited number of minor side-effects. Initial cluster of differentiation 20 (CD20)+ B cell depletion was seen in all patients. However, at 3 months, CD20+ B cells were starting to recover with five patients >35 cells/µl (range 35-152).(50) These data contrasts with previous work by Ruggenenti et al. using RTX given weekly (375 mg/m2) for 4 weeks. Pharmacokinetic (PK) analysis showed that RTX levels in this 2-dose regimen were 50% lower compared to non-proteinuric patients, which could potentially result in undertreatment.

Based on these results, the investigators recently conducted a study postulating that in patients with MN, 4 weekly doses of RTX would result in more effective B cell depletion, a higher remission rate and maintaining of the same safety profile compared to patients treated with RTX dosed at 1g x 2.

ELIGIBILITY:
Inclusion Criteria

* Idiopathic MN with diagnostic biopsy
* Female, must be post-menopausal, surgically sterile or practicing a medically approved method of contraception(no birth-control pill)
* Must be off prednisone or mycophenolate mofetil for >1 month and alkylating agents for >6 months.
* angiotensin-converting-enzyme inhibitor (ACEi) and/or Angiotensin II receptor blockers (ARB), for >3 months prior to randomization and adequate blood pressure (target BP <130/80 millimeter of mercury (mmHg) in >75% of the readings, but subjects with BP <140/80 mmHg in >75% of the readings will be eligible). Patients with documented evidence of >3 months treatment with maximal angiotensin II blockade, on an 3-hydroxy-3-methylglutaryl-CoA lyase (HMG-CoA) reductase inhibitor, and BP control (BP <140/80 mmHg in >75% of the readings) who remain with proteinuria >5g/24h may enter and be randomized to RTX/CSA without the need of the run-in/conservative phase of the study.
* Proteinuria >5g/24h on two 24-hour urine collection collected within 14 days of each other
* Estimated glomerular filtration rate (GFR) ≥40 ml/min/1.73m2 while taking ACEi/ARB therapy OR quantified endogenous creatinine clearance >40 ml/min/1.73m2 based on a 24-hour urine collection.

Exclusion Criteria

* Presence of active infection or a secondary cause of MN (e.g. hepatitis B, systemic lupus erythematosus (SLE), medications, malignancies). Testing for HIV, Hepatitis B and C should have occurred <2 years prior to enrollment into the study.
* Type 1 or 2 diabetes mellitus: to exclude proteinuria secondary to diabetic nephropathy. Patients who have recent history of steroid induced diabetes but no evidence on renal biopsy performed within 6 months of entry into the study are eligible for enrollment.
* Pregnancy or breast feeding for safety reasons
* History of resistance to CSA (or other calcineurin inhibitors, e.g. tacrolimus), RTX or alkylating agents (e.g. Cytoxan). Patients who previously responded to CSA/Calcineurin Inhibitor (CNI), RTX or alkylating agents with either a complete remission (CR) or partial remission (PR) but relapsed off CSA/CNI after 3 months or relapsed off RTX or alkylating agent after 6 months are eligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-11; Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C. Fervenza, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (21):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of Arizona, Tucson, Tucson, Arizona
  - Stanford University, San Francisco, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - New York University, New York, New York
  - Columbia University Medical Center, New York, New York
  - MetroHealth System (Case Western Reserve University), Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Froedtert Hospital, Milwaukee, Wisconsin
- Canada (3):
  - St. Paul's Hospital, Providence Health Care, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Centre hospitalier universitaire de Quebec - Hotel-Dieu de Quebec, Québec

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952
- [Derived] Xie J, Liu L, Mladkova N, Li Y, Ren H, Wang W, Cui Z, Lin L, Hu X, Yu X, Xu J, Liu G, Caliskan Y, Sidore C, Balderes O, Rosen RJ, Bodria M, Zanoni F, Zhang JY, Krithivasan P, Mehl K, Marasa M, Khan A, Ozay F, Canetta PA, Bomback AS, Appel GB, Sanna-Cherchi S, Sampson MG, Mariani LH, Perkowska-Ptasinska A, Durlik M, Mucha K, Moszczuk B, Foroncewicz B, Paczek L, Habura I, Ars E, Ballarin J, Mani LY, Vogt B, Ozturk S, Yildiz A, Seyahi N, Arikan H, Koc M, Basturk T, Karahan G, Akgul SU, Sever MS, Zhang D, Santoro D, Bonomini M, Londrino F, Gesualdo L, Reiterova J, Tesar V, Izzi C, Savoldi S, Spotti D, Marcantoni C, Messa P, Galliani M, Roccatello D, Granata S, Zaza G, Lugani F, Ghiggeri G, Pisani I, Allegri L, Sprangers B, Park JH, Cho B, Kim YS, Kim DK, Suzuki H, Amoroso A, Cattran DC, Fervenza FC, Pani A, Hamilton P, Harris S, Gupta S, Cheshire C, Dufek S, Issler N, Pepper RJ, Connolly J, Powis S, Bockenhauer D, Stanescu HC, Ashman N, Loos RJF, Kenny EE, Wuttke M, Eckardt KU, Kottgen A, Hofstra JM, Coenen MJH, Kiemeney LA, Akilesh S, Kretzler M, Beck LH, Stengel B, Debiec H, Ronco P, Wetzels JFM, Zoledziewska M, Cucca F, Ionita-Laza I, Lee H, Hoxha E, Stahl RAK, Brenchley P, Scolari F, Zhao MH, Gharavi AG, Kleta R, Chen N, Kiryluk K. The genetic architecture of membranous nephropathy and its potential to improve non-invasive diagnosis. Nat Commun. 2020 Mar 30;11(1):1600. doi: 10.1038/s41467-020-15383-w. PMID 32231244
- [Derived] Fervenza FC, Appel GB, Barbour SJ, Rovin BH, Lafayette RA, Aslam N, Jefferson JA, Gipson PE, Rizk DV, Sedor JR, Simon JF, McCarthy ET, Brenchley P, Sethi S, Avila-Casado C, Beanlands H, Lieske JC, Philibert D, Li T, Thomas LF, Green DF, Juncos LA, Beara-Lasic L, Blumenthal SS, Sussman AN, Erickson SB, Hladunewich M, Canetta PA, Hebert LA, Leung N, Radhakrishnan J, Reich HN, Parikh SV, Gipson DS, Lee DK, da Costa BR, Juni P, Cattran DC; MENTOR Investigators. Rituximab or Cyclosporine in the Treatment of Membranous Nephropathy. N Engl J Med. 2019 Jul 4;381(1):36-46. doi: 10.1056/NEJMoa1814427. PMID 31269364
- [Derived] Fervenza FC, Canetta PA, Barbour SJ, Lafayette RA, Rovin BH, Aslam N, Hladunewich MA, Irazabal MV, Sethi S, Gipson DS, Reich HN, Brenchley P, Kretzler M, Radhakrishnan J, Hebert LA, Gipson PE, Thomas LF, McCarthy ET, Appel GB, Jefferson JA, Eirin A, Lieske JC, Hogan MC, Greene EL, Dillon JJ, Leung N, Sedor JR, Rizk DV, Blumenthal SS, Lasic LB, Juncos LA, Green DF, Simon J, Sussman AN, Philibert D, Cattran DC; Mentor Consortium group. A Multicenter Randomized Controlled Trial of Rituximab versus Cyclosporine in the Treatment of Idiopathic Membranous Nephropathy (MENTOR). Nephron. 2015;130(3):159-68. doi: 10.1159/000430849. Epub 2015 Jun 12. PMID 26087670
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Treatment Arm: Patients randomized to the RTX arm will receive 1000 mg IV on Days 1 and 15. Patients who achieve complete remission at 6 months will not be retreated. A second course of RTX 1000 mg IV will be administered at study month 6 for individuals who have not achieved a complete remission, but have achieved a minimum of >25% reduction in Time 0 proteinuria. Dosing at study month 6 will be independent of CD19+ B cell count.
  Rituximab: 1000 mg, I.V. on Days 1 and 15 and will be retreated at month 6 independent of CD19+ B cell count
Period: Overall Study
Arm/Group | Rituximab Treatment Arm | Cyclosporine Treatment Arm
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab Treatment Arm | Cyclosporine Treatment Arm | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.6) | 52.2 (12.4) | 52.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 47 | 53 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 11 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 51 | 49 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Remission Status
Description: The number of subjects to reach the composite of maintaining complete remission or partial remission at 24 months after randomization will be the primary endpoint.
Time Frame: 24 months after randomization
Measure: Count of Participants; unit: Participants
Groups:
- Rituximab Treatment Arm: Patients randomized to the Rituximab (RTX) arm will receive 1000 mg IV on Days 1 and 15. Patients who achieve complete remission at 6 months will not be retreated. A second course of RTX 1000 mg IV will be administered at study month 6 for individuals who have not achieved a complete remission, but have achieved a minimum of >25% reduction in Time 0 proteinuria. Dosing at study month 6 will be independent of Cluster of Differentiation 19 (CD19)+ B cell count.
  Rituximab: 1000 mg, I.V. on Days 1 and 15 and will be retreated at month 6 independent of CD19+ B cell count
- Cyclosporine Treatment Arm: Patients randomized to the Cyclosporine (CsA) arm will be started at a dose of CsA = 3.5 mg/kg/day p.o. divided into 2 equal doses given at 12 hour intervals. Target trough CsA blood levels are 125 to 175 ng/ml. Patients will have their doses adjusted according to their blood levels of CSA as monitored every 2 weeks until the target trough level is reached. If a complete remission is achieved by 6 months, CSA will be tapered and discontinued over a three-month period. If after 6 months there has not been a reduction in proteinuria of at least 25% of baseline values, the drug will also be discontinued. If there has been a >25% reduction in baseline proteinuria (but not complete remission) the CSA will be continued for an additional 6 months.
Arm/Group | Rituximab Treatment Arm | Cyclosporine Treatment Arm
Number analyzed (Participants) | 65 | 65
Participants | 39 | 13
Statistical Analysis 1: Comparison: Rituximab Treatment Arm vs Cyclosporine Treatment Arm; Test type: Superiority; p = 0.001, Chi-squared; Risk Difference (RD) = 40, 95% CI 2-sided [24.6 to 55.4]

2. Secondary Outcome: Remission Status
Description: The number of subjects to reach either complete remission or partial remission at 12 months after randomization.
Time Frame: 12 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab Treatment Arm | Cyclosporine Treatment Arm
Number analyzed (Participants) | 65 | 65
Participants | 39 | 34
Statistical Analysis 1: Comparison: Rituximab Treatment Arm vs Cyclosporine Treatment Arm; Test type: Non-Inferiority — With a non-inferiority margin of 15%. enrollment of 63 evaluable patients per study are is required to achieve 80% power to show that RTX is not inferior; p = 0.009, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from enrollment through month 18, for each subject, approximately 18 months total.
Arm/Group | Rituximab Treatment Arm | Cyclosporine Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 11/65 | 20/65
Other Adverse Events (participants affected / at risk) | 46/65 | 51/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Treatment Arm (N=65) | Cyclosporine Treatment Arm (N=65)
Benign neoplasms (General disorders) | 1 (1) | 0 (0)
Blood and lymphatic system (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiovascular (Cardiac disorders) | 1 (1) | 7 (7)
Endocrine or metabolic (Endocrine disorders) | 2 (2) | 1 (1)
General (General disorders) | 1 (1) | 0 (0)
Infections (Infections and infestations) | 4 (5) | 8 (8)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Nervous system (Nervous system disorders) | 1 (1) | 1 (1)
Renal and urinary (Renal and urinary disorders) | 0 (0) | 2 (2)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Treatment Arm (N=65) | Cyclosporine Treatment Arm (N=65)
Benign neoplasms (General disorders) | 1 (1) | 1 (1)
Blood and lymphatic system (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Cardiovascular (Cardiac disorders) | 5 (6) | 11 (14)
Ear (Ear and labyrinth disorders) | 3 (3) | 1 (2)
Endocrine or metabolic (Endocrine disorders) | 7 (9) | 6 (15)
Eye (Eye disorders) | 1 (1) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 7 (11) | 18 (34)
General (General disorders) | 25 (42) | 15 (24)
Immune system (Immune system disorders) | 1 (1) | 1 (1)
Infections (Infections and infestations) | 17 (28) | 20 (26)
Injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 10 (17) | 18 (27)
Nervous system (Nervous system disorders) | 11 (15) | 16 (26)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Psychiatric (Psychiatric disorders) | 1 (1) | 5 (7)
Renal and Urinary (Renal and urinary disorders) | 6 (8) | 16 (19)
Reproductive system and breast (Reproductive system and breast disorders) | 3 (4) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 6 (11)
Skin (Skin and subcutaneous tissue disorders) | 12 (14) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT01180036/Prot_SAP_000.pdf